CLINICAL TRIAL: NCT03825471
Title: Effects of Cranial Electrotherapy Stimulation on Anesthetics Consumption, Perioperative Cytokines Response, and Postoperative Pain in Patients Undergoing Colonic Surgery
Brief Title: Cranial Electrotherapy Stimulation on Anesthetics Consumption and Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yi-hsuan Huang, Attending Physician, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CES and Postoperative pain
Record Dates: First submitted 2019-01-22; First posted 2019-01-31 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Opioid Use; Cytokine
Keywords: Cranial electrotherapy stimulation (CES); Autonomic nervous system; acute postoperative pain; colon cancer surgery; patient-controlled analgesia (PCA)
MeSH Terms: conditions — Pain, Postoperative | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- electrotherapy (Experimental): Patients undergoing CES and general anesthesia in colon cancer surgery
  Interventions: Procedure: electrotherapy; Drug: Opioid Anesthetics; Procedure: colon cancer surgery
- Opioid Anesthetics (Placebo Comparator): Patients undergoing general anesthesia in colon cancer surgery
  Interventions: Procedure: electrotherapy; Drug: Opioid Anesthetics; Procedure: colon cancer surgery

INTERVENTIONS:
Procedure: electrotherapy — Cranial electrotherapy stimulation
Drug: Opioid Anesthetics — consumption of opioids during general anesthesia
  Other Names: Opioid consumption during general anesthesia
Procedure: colon cancer surgery — laparoscopic colon cancer surgery

SUMMARY:
Cranial electrotherapy stimulation (CES) is a non-invasive intervention to treat anxiety, depression, insomnia, and pain. But clinical studies and applications of CES in relation to acute postoperative pain are few. tThe investigators investigate a double-blind, randomized controlled trial to figure out if intraoperative CES could decrease dosage of intraoperative anesthetics and patient-controlled analgesia (PCA) consumption in patients undergoing colon cancer surgery.

DETAILED DESCRIPTION:
Cranial electrotherapy stimulation (CES) is a non-invasive and safe intervention, transmitting microcurrents of brain stimulation and releasing various neurotransmitters such as endorphin and downstream hormones to modulate autonomic nervous system, as a result, for treating anxiety, depression, insomnia, and pain.

Acute postoperative pain annoys patients receiving surgery. Once acute postoperative pain is poorly controlled, it may result in adverse acute effects (i.e., physiologic and psychologic stress), chronic effects (i.e., delayed long-term recovery and chronic pain), and, in consequence, excess length of hospitalization and extra costs. Besides, inflammatory reactions mediated by immune system are formed after tissue injury (e.g. trauma, surgery, etc), release serial inflammatory cytokines and are related to pain signal transmission. However, clinical studies and applications of CES focus on management of chronic pain, modulation of mood and insomnia rather than acute postoperative pain in recent years.

The investigators investigate a double-blind, randomized controlled trial to figure out if intraoperative CES could decrease dosage of intraoperative anesthetics and patient-controlled analgesia (PCA) consumption in patients undergoing colon cancer surgery. The investigators also collect blood samples before and after surgery for analysis of serum cytokines. Meanwhile, Bispectral IndexTM (BISTM) monitoring and Analgesia Nociception Index (ANI) are prescribed during the surgery not only for measuring of the effects of anesthetics and sedatives on the brain, but also evaluating perioperative analgesia. Thereby, the effectiveness of CES for management of acute postoperative pain may introduce clinicians for alternative application of pain control after surgery in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colon cancer surgery

Exclusion Criteria:

* presence of an implantable device (e.g., pacemaker)
* pregnancy
* having a known mental illness (e.g., schizophrenia, mood disorder, bipolar disorder, etc.
* cancer of the head and neck or brain tumor or brain metastasis
* having delirium

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
dosage of intraoperative anesthetics | during surgery
  The consumption of total amount of supplemental analgesics administered during colon cancer surgery
Rescue analgesics | from the end of the surgery to postoperative 72 hours
  The consumption of total amount of rescue analgesics administered after colon cancer surgery
Differences in Pain Intensity Between CES intervention and the control group | from the end of the surgery to postoperative 72 hours
  Pain assessment of NRS pain intensity scores and patient satisfaction assessed by the NRS through end of surgery to postoperative 72 hours

SECONDARY OUTCOMES:
dosage of patient-controlled analgesia (PCA) consumption | from the end of the surgery to postoperative 72 hours
  postoperative PCA consumption
serum concentration of serum cytokine | from the beginning of the surgery to postoperative 72 hours
  proinflammatory and antiinflammatory cytokines (IL-1a, IL-2, IL-6, IL-7, TNF-a, IL-4, IL-10, IL-10, IL-1, TGF-b)
Number of Participants with CES and control groups | during surgery
  patient characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Yi-hsuan Huang, MD, Principal Investigator — TriService General Hospital
Locations (1):
- TriService General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee SH, Kim WY, Lee CH, Min TJ, Lee YS, Kim JH, Park YC. Effects of cranial electrotherapy stimulation on preoperative anxiety, pain and endocrine response. J Int Med Res. 2013 Dec;41(6):1788-95. doi: 10.1177/0300060513500749. PMID 24265330